CLINICAL TRIAL: NCT01538394
Title: Randomized Double-blind Trial of Two Parallel Groups Design to Evaluate the Efficacy of Smoking Cessation With Combined (Varenicline Plus Nicotine Patches) Versus Monotherapy (Varenicline Plus Placebo Patches)
Brief Title: Clinical Trial to Evaluate the Efficacy of Smoking Cessation
Acronym: COMBIVAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Josep Maria Ramon Torrell, PhD (Other)
Responsible Party: Sponsor-Investigator, Josep Maria Ramon Torrell, PhD, Josep Maria Ramon Torrell, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: VAR/01/011
Record Dates: First submitted 2012-02-14; First posted 2012-02-24 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; abstinence; clinical trial; varenicline; nicotine
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline & nicotine patches (Experimental): Combined therapy by using Varenicline plus nicotine patches.The intervention-phase will comprise two fasses:
  * Pre-NRT: Patients take 1 week VRN impregnation (0.5mg/day during the first 3 days + 0.5mg twice daily for the next for days)
  * Treatment: starting at day 8 and during the next 11 weeks patients continue taking VRN 1mg twice daily plus placebo transdermal patches of 30cm2/24 hours per 8 weeks and then 20cm2/24 hours per 3 weeks.
  Interventions: Drug: Varenicline; Drug: Nicotine patches
- Varenicline & placebo patches (Placebo Comparator): Monotherapy by using Varenicline plus placebo patches.The intervention-phase will comprise two fasses:
  * Pre-NRT: Patients take 1 week VRN impregnation (0.5mg/day during the first 3 days + 0.5mg twice daily for the next for days)
  * Treatment: starting at day 8 and during the next 11 weeks patients continue taking VRN 1mg twice daily plus nicotine transdermal patches of 30cm2/24 hours per 8 weeks and then 20cm2/24 hours per 3 weeks.
  Interventions: Drug: Varenicline; Drug: Placebo (nicotine patches)

INTERVENTIONS:
Drug: Varenicline
  Other Names: champix
Drug: Nicotine patches
  Other Names: Campix; Nicotinell
  Arms: Varenicline & nicotine patches
Drug: Placebo (nicotine patches)
  Arms: Varenicline & placebo patches

SUMMARY:
The purpose of this study is to assess the efficacy of smoking cessation by using varenicline as monotherapy (VRN + placebo patches) or combined therapy (VRN + nicotine patches).

DETAILED DESCRIPTION:
Seven first-line pharmacotherapies are currently available and recommended by clinical practice guidelines for treating tobacco dependence, all of them have been proven to be effective for increasing tobacco abstinence rates when used as monotherapy. However, not all smokers are able to quit with monotherapy. Some smokers may benefit from combination therapy that includes the simultaneous use of different nicotine replacement therapies (NRTs) or medications with different mechanisms of action (e.g. NRT and bupropion). Combination therapy with different drugs may provide a therapeutic advantage by increasing serum nicotine concentrations, and may capitalize on synergy obtained from two different mechanisms of action. This is why controversy exists regarding this approach as the cost effectiveness of this approach has not been clearly demonstrated neither if the genetic profile determine different treatment responses.

Data from a varenicline pharmacokinetic study have documented that among smokers not instructed to quit and who continued smoking during treatment , varenicline was associated with a 60-80 % of reduction of number of cigarettes and, on the other hand, with a diminution of plasmatic nicotine and cotinine concentrations. (See some studies and trials in the Background Information).

This , led to hypotheses that : a) varenicline not saturate completely all acetylcholinergic receptors with a incomplete response and ; b) varenicline replace incompletely the dopaminergic effect of smoking, with continuous craving. The investigators considered that some smokers may need NRT in addition to varenicline to reduce withdrawal and cravings to smoke.

Finally, available data suggests that combination therapy may increase abstinence rates compared with monotherapy [OR: 2.4 (2.1- 2.7)] without a significant increase of adverse events. So the periodicity, regimen/dose, and periods of combined treatment may be considered as safe as the monotherapy even in an off-label indication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years old
* Smoking 20 or more cigarettes per day
* Wants to stop smoking(seeking treatment)
* No period of smoking abstinence longer than 3 months in the past year
* Be able to give informed consent to participate
* Complete the study questionnaires
* Female smokers will be eligible providing they are not breastfeeding, pregnant (negative pregnancy test) or at risk of becoming pregnant

Exclusion Criteria:

* Previous use of nicotine transdermal patches or varenicline (VRN) in the last 6 months
* Cigar, pipe and oral tobacco users who do not smoke 20 or more cigarettes per day
* Those who meet the criteria contra-indicating nicotine patches or VRN use, as described in the Summaries Product Characteristics
* Those with previous severe adverse reactions to nicotine patch or to VRN
* Those currently taking either medication for smoking cessation that they are unwilling to stop or taking medication with a known influence on smoking cessation that they should not stop (e.g. nortriptyline for depression)
* Those who are non-Spanish neither Catalan speakers
* Those deemed unsuitable for the study by their smoking cessation physicians; -- Unstable diseases within the previous 6 months
* Diagnoses of or treatment for major depression last 6 months or psychotic disorder; or drug or alcohol dependence within the previous 12 months
* Skin disorders that cause a difficulty of nicotine absorption by patches as Psoriases as well as general dermatitis
* Clinically significant renal or hepatic impairment or dysfunction
* Pregnant or breast-feeding women
* women who do not use neither want to use any effective anticonceptive method.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of combined therapy (VRN+nicotine patches) versus monotherapy (VRN+placebo patches) in smoking cessation assessed as continuous abstinence rate (CAR) from week 2 to week 12. | Participants will be followed for the duration of treatment, 12 weeks.
  The primary endpoint will be the continuous abstinence rate (CAR) from week 2 (w2) to week 12 (w12) measured objectively during the treatment phase by the CO exhaled.

SECONDARY OUTCOMES:
i) Determine safety of combined therapy (VRN+nicotine patches) versus monotherapy (VRN+placebo patches) | Every two weeks from week 2 to 12
  The secondary endpoints will be related to efficacy [continued abstinence rate (CAR) from week 2 to week 52, (CAR) from week 2 to week 6, (CAR) from week 2 to week 24, (CAR) from week 2 to week 36; point abstinence rate (PAR) at week 6, PAR at week 12, PAR at week 24, PAR at week 36, PAR at week 52], safety and cravings appearances.

CONTACTS AND LOCATIONS:
Overall Officials: JOSEP M RAMON TORRELL, PhD, Study Director — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Ramon JM, Morchon S, Baena A, Masuet-Aumatell C. Combining varenicline and nicotine patches: a randomized controlled trial study in smoking cessation. BMC Med. 2014 Oct 8;12:172. doi: 10.1186/s12916-014-0172-8. PMID 25296623